CLINICAL TRIAL: NCT06829238
Title: Assessment of Metformin for Restoration of Immune Homeostasis in HIV+ and HIV- Individuals With a History of Injection Drug Use (MET-IH)
Brief Title: Assessment of Metformin for Restoration of Immune Homeostasis in HIV+ and HIV- Individuals With a History of Injection Drug Use
Acronym: (MET-IH)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Ellen Eaton, Dr. Ellen Eaton, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000543853; 1R01DA060692-01A1 (NIH)
Record Dates: First submitted 2025-02-04; First posted 2025-02-17 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Systemic Inflammation; Immune Dysregulation; Injection Drug Use; HIV
Keywords: Metformin; Immune restoration; Vaccine response; People who inject drugs (PWID)
MeSH Terms: interventions — Metformin; smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin Group (Experimental): Participants will receive Metformin ER (500mg increasing to 1000mg) for 16 weeks to assess immune restoration and inflammatory response.
  Interventions: Drug: Metformin; Biological: Jynneos; Biological: Capvaxvie
- Placebo Group (Placebo Comparator): Control Group
  Interventions: Drug: Placebo; Biological: Jynneos; Biological: Capvaxvie

INTERVENTIONS:
Drug: Metformin — Participants will receive Metformin ER (500mg increasing to 1000mg) or placebo for 16 weeks to assess immune restoration and inflammatory response.
  Arms: Metformin Group
Drug: Placebo — Participants will receive placebo for 16 weeks and assess immune restoration and inflammatory response.
  Arms: Placebo Group
Biological: Jynneos — All participants will take a Jynneos (MPOX) vaccine.
Biological: Capvaxvie — All participants will take a Capvaxvie (PCV21, pneumococcal) vaccine.

SUMMARY:
This randomized clinical trial (RCT) evaluates whether metformin can reduce systemic inflammation and improve immune function in individuals with a history of injection drug use, with or without HIV. Participants will receive metformin or placebo and undergo immune system assessments, including vaccine response evaluations.

DETAILED DESCRIPTION:
The study aims to assess the impact of metformin on immune dysregulation among 100 adults (ages 18-64) with a history of injection drug use. Participants will be randomized 1:1 to metformin (500mg increasing to 1000mg) or placebo for 16 weeks, during which they will receive Jynneos (MPOX) and Capvaxvie (PCV21, pneumococcal) vaccines. Immunologic responses will be monitored over 6 months post-enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent.
* Stated willingness to comply with all study procedures and availability for the study duration.
* Aged 18 to 64 years old.
* Weight of at least 110 lbs.
* Body Mass Index (BMI) of 18.5-40. Enrollment of individuals with BMI >40, deemed in good health, may be considered with approval.
* Willingness to receive Jynneos (MPOX) and Capvaxvie vaccines.
* Ability to take oral medication and willingness to adhere to the metformin treatment regimen.
* History of injection opioid, amphetamine, and/or cocaine use within the past 10 years (self-report).
* Use of non-prescription opioid, amphetamine, and/or cocaine within the past 30 days (self-report).
* Clinically confirmed urine drug screen for opioid, amphetamine, and/or cocaine within the past 30 days.
* Serum CRP > 3 mg/dL.
* Glucose level between 70-180 mg/dL (non-fasting).
* Hemoglobin A1c (HbA1c) of 5.0-6.4%.
* CD4 count > 200 cells/ml.
* If HIV-positive, HIV viral load < 200 copies/ml.
* If HIV-positive, on anti-retroviral therapy (ART) for >12 months.

Exclusion Criteria:

* Inability to give informed consent.
* Refusal or inability to have blood drawn.
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, platelet disorder requiring precautions).
* Pregnant or nursing individuals.
* Diabetes mellitus.
* History of severe renal impairment or eGFR <60 mL/min/1.73m².
* Creatinine clearance <60 mL/min.
* History of liver disease.
* ALT/AST > 3× the upper limit of normal.
* Total bilirubin >1.4 mg/dL.
* Albumin <3.5 g/dL.
* Prothrombin >1.5× the upper limit of normal.
* AUDIT-C score ≥8.
* Hemoglobin <9.0 g/L.
* Absolute neutrophil count <1,000/mL.
* Platelet count <100,000/mL.
* History of acute or chronic metabolic acidosis.
* Serum bicarbonate <22 mEq/L.
* Anion gap >10 mEq/L.
* Serum lactate >2.2 mmol/L.
* Serum vitamin B12 <250 pg/mL.
* History of chronic diarrhea.
* Current use of metformin or other diabetes medications.
* History of myocardial infarction, endocarditis, stroke, heart failure, chronic obstructive pulmonary disease, or sepsis.
* Use of medications such as furosemide, nifedipine, ranolazine, vandetanib, or cimetidine (current or within the past 30 days).
* Active hepatitis B infection.
* Hepatitis C infection within 6 months of study entry; individuals with prior hepatitis C must be at least 6 months post-treatment with direct-acting antivirals.
* Previous receipt of Jynneos or pneumococcal vaccine within the past two years (self-report).
* Severe allergic reaction to metformin, Jynneos, or Capvaxvie (self-report). Blood donations exceeding 450 mL in the 8 weeks prior to enrollment, accounting for study-related blood draws.
* Any medical, psychiatric, social condition, or responsibility that, in the investigator's judgment, could interfere with study procedures.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Serum C-reactive Protein (CRP) | Baseline to Week 16
  Assessed by Enzyme Linked Immunosorbent Assay (ELISA) of blood samples collected at baseline and at 16 weeks. Reported in mg/dL.

SECONDARY OUTCOMES:
Change in exhausted B cells | Baseline to Week 16
  Assessed by flow cytometry of blood samples collected at baseline and at 16 weeks. Reported as percentage of total B cells.
Change in exhausted T cells | Baseline to Week 16
  Assessed by flow cytometry of blood samples collected at baseline and at 16 weeks. Reported as percentage of total T cells.
Change in MPOX vaccine-specific IgG antibody. | Baseline to Week 13
  Assessed by Enzyme Linked Immunosorbent Assay (ELISA) of blood samples collected at baseline and at 13 weeks. Reported as micrograms/mL.
Change in PCV21 vaccine-specific IgG antibody. | Baseline to Week 9
  Assessed by Enzyme Linked Immunosorbent Assay (ELISA) of blood samples collected at baseline and at 9 weeks. Reported as micrograms/mL.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided